CLINICAL TRIAL: NCT04832893
Title: Effects of Different Masks on Metabolic Parameters, Inspiratory Muscle Strength and Perceived Effort During Low Intensity Aerobic Exercise
Brief Title: Use of Masks on Metabolic Parameters and Inspiratory Muscle Strength During Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UFV_20/2021
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Use of FFP2 respirator (Active Comparator): Using of FFP2 respirator during the 30 minutes test
  Interventions: Diagnostic Test: steady intensity aerobic test of 30 minutes long
- Use of surgical mask (Active Comparator): Using of surgical mask during the 30 minutes test
  Interventions: Diagnostic Test: steady intensity aerobic test of 30 minutes long
- no mask (Sham Comparator): The 30 minutes test will be carried out without mask
  Interventions: Diagnostic Test: steady intensity aerobic test of 30 minutes long

INTERVENTIONS:
Diagnostic Test: steady intensity aerobic test of 30 minutes long — the use of different type of masks during an aerobic exercise

SUMMARY:
The purpose of this study will be to assess the effects of the use of masks on inspiratory muscle strength, metabolic parameters, heart rate, subjective perception of effort and the sensation of dyspnea before, during and after an aerobic test of 30 minutes long and a fixed load at lactate threshold. A randomized study of repeated measures will be carried out. A total sample of 35 active participants will be recruited. All participants will carried out a lactate threshold test and then 3 visits to the laboratory (separated at least 48 hours from each other) in order to perform 3 test of 30 minutes long without mask, with a surgical mask or with a FFP2 respirator (in a randomized order) at an intensity around lactate threshold intensity. Maximal inspiratory pressure, oxygen saturation, heart rate, blood lactate concentration, subjective perception of effort and dyspnea will be assessed before, during and after the 3 fixed intensity tests.

ELIGIBILITY:
Inclusion Criteria:

* carrying out at least 2 days of physical activity per week

Exclusion Criteria:

* cardiac disease
* pulmonary disease
* chronic inflammatory disease
* sedentary behaviour

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | change from baseline inspiratory muscle strength after the 30 minutes test
  Inspiratory muscle strength will be measured in mmHg with a Power-breathe device

SECONDARY OUTCOMES:
lactate concentrations | change from baseline after 10 minutes, 20 minutes and 30 minutes during the test
  lactate concentration will be measured in mmol/L with a Lactate Pro 2 device
oxygen saturation | change from baseline after 10 minutes, 20 minutes and 30 minutes during the test
  oxygen saturation will be measured in %
heart rate | change from baseline after 10 minutes, 20 minutes and 30 minutes during the test
  heart rate will be measured in beats per minute with a polar H10 device
rate of perceived effort | change from baseline after 10 minutes, 20 minutes and 30 minutes during the test
  rate of perceived effort will be obtained through the Borg´ scale
sensation of dyspnea | change from baseline after 10 minutes, 20 minutes and 30 minutes during the test
  sensation of dyspnea will be obtained through a visual analog scale from 0 to 10 points

CONTACTS AND LOCATIONS:
Overall Officials: Davinia Vicente Campos, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No